CLINICAL TRIAL: NCT01716897
Title: A Randomized, Open-label, 3-treatment Crossover Study to Determine the Bioavailability of E2609 Tablets Compared to Capsules and the Effect of Food on Absorption in Healthy Caucasian Male Adults
Brief Title: An Study to Determine the Bioavailability of E2609 Tablets Compared to Capsules and the Effect of Food on Absorption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E2609-A001-007
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50 mg E2609 capsule formulation in fasted state (Other): 50 mg E2609 capsule formulation
  Interventions: Drug: E2609
- 50 mg E2609 tablet formulation in fasted state (Other): 50 mg E2609 tablet formulation in fasted state
  Interventions: Drug: E2609
- 50 mg tablet formulation in fed state (Other): 50 mg E2609 tablet formulation in fed state
  Interventions: Drug: E2609

INTERVENTIONS:
Drug: E2609

SUMMARY:
This study will be a single-center, open-label, randomized, 3-treatment crossover study of single oral doses of an API-capsule formulation of E2609 under fasted conditions and a tablet formulation administered under fed and fasted conditions in healthy subjects.

ELIGIBILITY:
Inclusion Criteria

1. Caucasian males defined as persons of a European or Latin American descent
2. Healthy male 30 to 55 years inclusive at the time of informed consent
3. Body mass index (BMI) of 18 to 32 kg/m2 at Screening
4. Subjects must have had a successful vasectomy (confirmed azoospermia), or they and their female partners must not be of childbearing potential or must be practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation. No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.

Exclusion Criteria

1. Any history of seizures or epilepsy (not including a history of simple febrile seizures in childhood) or disturbance of consciousness likely to be due to seizures
2. Any medical condition which, in the opinion of the investigator has high risk of seizures (e.g., history of traumatic brain injury associated with loss of consciousness or amnesia, alcohol abuse, substance abuse) at Screening or within past 5 years
3. Any history of cerebrovascular disease (stroke or transient ischemic attack)
4. A history of prolonged QT/QTc interval or prolonged period from the beginning of the QRS complex to the end of the T wave on an ECG (QT)/ QT corrected for heart rate using Fridericia?s formula (QTcF) interval (QTcF > 450 ms) as demonstrated by the mean of triplicate electrocardiogram (ECGs) (recorded at least 1 min apart) at Screening or Baseline Period
5. Any other clinically significant ECG abnormalities at Screening or Baseline Periods, e.g. component of the ECG cycle from onset of atrial depolarization to onset of ventricular depolarization (PR)>220 ms, component of ECG wave representing ventricular depolarization (QRS)>110 ms
6. Hypersensitivity to the study drugs or any of their excipients

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
AUC(0-inf) ratio, new tablet vs. capsule | 0 -144 hours
AUC(0-inf) ratio, fed state vs. fasted state, both after administration of new tablet | 0 - 144 hours
Cmax ratio, new tablet vs. capsule | 0 - 144 hours
Cmax ratio, fed state vs. fasted state, both after administration of new tablet | 0 - 144 hours

SECONDARY OUTCOMES:
incidence of Adverse events | 5.5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Haykop Gevorkyan, Principal Investigator — California Clinical Trials Medical Group/Parexel
Locations (1):
- California Clinical Trials/Parexel, Glendale, California, United States